CLINICAL TRIAL: NCT00691704
Title: Lenalidomide and Low Dose Dexamethasone Induction Therapy Followed by Low Dose Melphalan, Prednisone, Lenalidomide and Bortezomib Sequential Maintenance Therapy for Newly Diagnosed High-risk Multiple Myeloma
Brief Title: Celgene High Risk Multiple Myeloma (MM) Revlimid Induction and Maintenance Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cristina Gasparetto (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Cristina Gasparetto, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00002869
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Bortezomib; Melphalan; Prednisone; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High-risk Multiple Myeloma (Experimental): Lenalidomide Induction (with Low Dose Dexamethasone) Therapy Followed by Low Dose Melphalan, Prednisone, Lenalidomide and Bortezomib Sequential Maintenance Therapy
  Interventions: Drug: Lenalidomide Induction; Drug: Sequential Maintenance Therapy

INTERVENTIONS:
Drug: Lenalidomide Induction — Induction: Lenalidomide 25 mg daily on Days 1-21 followed by 7 day rest and Dexamethasone 40 mg by mouth (po) daily on Days 1, 8, 15 and 22 every 28 days for 4 cycles.
  Other Names: Lenalidomide
Drug: Sequential Maintenance Therapy — Subjects who achieve >partial response (PR) following induction therapy will receive repeating triplet cycles of alternating low dose therapy until progression, poor tolerance or toxicity. Subjects who complete 24 months of maintenance will be removed from study unless they achieved > stable disease (SD) from maintenance (per discussion with physician):
  * 325 mg aspirin for deep vein thrombosis (DVT) prophylaxis
  * Cycle 1, 4, 7, etc. - bortezomib 1.3 mg/m2 on day 1 and 8 of a 28-day cycle
  * Cycle 2, 5, 8 etc. - Melphalan 6 mg/m2 by mouth (po) daily on Days 1-7
  * Prednisone 60 mg /m2 po daily on Days 1-7 of a 28-day cycle
  * Cycle 3, 6, 9, etc. Lenalidomide 10 mg po daily on Days 1-21 of a 28 day cycle.
  Other Names: Lenalidomide (Revlimid); Bortezomib (Velcade); Melphalan; Prednisone; Aspirin

SUMMARY:
The purpose of this study is to evaluate the effectiveness of induction therapy with lenalidomide and low dose dexamethasone followed by sequential low dose bortezomib followed by low dose Melphalan and Prednisone, then followed by low dose lenalidomide for multiple cycles in subjects with high risk Multiple Myeloma (MM). The primary objective is to evaluate the efficacy as measured by the progression free survival (PFS) at 2 years of low dose sequential therapy following four cycles of induction therapy with lenalidomide/low-dose dexamethasone in subjects with symptomatic high risk multiple myeloma, who have received no prior treatment. A total of 35 subjects were estimated to be accrued to this Phase II trial over a period of subjects who are still progression-free at 2 years. Two years will be as measured from date of registration to the trial. Progression will include disease progression (DP) as well as death due to any cause. Data will be analyzed and reported by the PI after 1 and 2 years of initiation of the study. All subsequent data collected may be analyzed and reported in a follow-up clinical report. The PI and independent reviewers will meet to review the efficacy and safety data and determine a risk/benefit analysis in this subject population.

DETAILED DESCRIPTION:
Study design: A total of 35 subjects who were newly diagnosed, high risk Multiple Myeloma (high risk defined by the presence of one or more of the following: t(4;14), t(14;16), deletion of 17p13 (p53) by FISH, deletion of chromosome 13 or aneuploidy on metaphase analysis) were estimated to be accrued to this Phase II trial over a period of about 3 years.

The primary objective is to estimate the proportion of subjects who are still progression-free at 2 years. Two years is measured from date of registration to the trial. Progression will include disease progression as well as death due to any cause. Time to response, defined only for the responders, is defined as the time from the date of initiation of treatment to the first documentation of a confirmed response. Duration of response among subjects achieving a sustained complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR) will be defined as the length of the interval from initial PR to time of disease progression. Progression free survival (PFS) is defined for all subjects as the time from the date of initiation of treatment to the date of first documentation of relapse, progression, or death due to any cause. Time to progression (TTP) is defined for all subjects as the time from initiation of treatment to disease progression with deaths owing to causes other than progression not counted as events, but censored (Durie et al., 2006). Overall survival (OS) is defined as the time from the date of initiation of treatment to the date of death due to any cause. The Garban et al. trial found a 2-year progression-free rate of about 0.60 in 212 similar subjects. If a 2-year rate of 0.60 were to be observed in this trial, we would consider the treatment a success. A rate of 0.60 has an exact 80% confidence interval (CI) of 0.48 - 0.71.

True 2-year Probability of observing Progression-free a rate ≥ 0.60 0.48 0.11 0.52 0.22 0.56 0.38 0.60 0.57 0.64 0.75 0.68 0.88 0.72 0.95

DOSING REGIMEN(S):

Induction therapy: Lenalidomide 25 mg daily on Days 1-21 followed by 7 day rest and Dexamethasone 40 mg by mouth (po) daily on Days 1, 8, 15 and 22 every 28 days for 4 cycles. Subjects will receive 325 mg aspirin for deep vein thrombosis (DVT) prophylaxis.

Following induction therapy: Stem cell collection and cryopreservation - Subjects who achieve sCR, CR,VGPR and PR, are eligible for future stem cell transplant procedure.

Maintenance sequential therapy - Subjects who achieve >PR following induction therapy will receive repeating triplet cycles of alternating low dose therapy:

* Subjects will receive 325 mg aspirin for DVT prophylaxis.
* Cycle 1, 4, 7, etc - bortezomib 1.3 mg/m2 on day 1 and 8 of a 28-day cycle
* Cycle 2, 5, 8 etc- Melphalan 6 mg/m2 po daily on Days 1-7 days and Prednisone 60 mg/m2 po daily on Days 1-7 of a 28-day cycle
* Cycle 3, 6, 9, etc. Lenalidomide 10 mg po daily on Days 1-21 of a 28 day cycle.

Subjects will continue sequential alternating triplet cycles until time of progression or discontinuation due to poor tolerance or toxicity. Subjects who complete 24 months of maintenance therapy will be removed from study. Subjects who have achieved > stable disease (SD) from maintenance may continue for longer than 24 months after discussion with their physicians.

Efficacy/response assessments (including skeletal survey, quantification of M-protein, immunoglobulins, bone marrow aspiration, biopsy & morphology, serum free-light chain assay, and immunofixation of serum & urine) are scheduled to occur within 7 days after completion of Cycle 2 and 4 during induction and then every third cycle during maintenance starting at the end of Cycle 3 (+/- 14 days). Efficacy assessments will also be done at discontinuation.

Subjects will be assessed for disease response according to the modified and updated European Group for Blood and Bone marrow Transplant (EBMT) criteria (Durie 2006, Blade 1998). Response categories are listed in Appendix 15.3.

Data from all subjects who receive any study drug will be included in the safety analyses. Subjects who entered the study and did not take any of the study drug and had this confirmed, will not be evaluated for safety. The severity of the toxicities will be graded according to the National Cancer Institute's (NCI) common terminology criteria for adverse events (CTCAE) v3.0. Safety evaluation will be based on the incidence, intensity and type of adverse events: Karnofsky performance score (KPS) and clinically significant changes in the subject's physical examination findings, vital sign measurements, and clinical laboratory results. Exposure to study drug and reasons for discontinuation of study treatment will be tabulated.

Analyses: The proportion of subjects progression-free at the times of full restaging (i.e., at 6, 12, 18, 24, 36 months) will be calculated with 80% confidence intervals and descriptively compared to the rates in the Garban et al. paper. Time-to-progression (TTP) will be estimated with the Kaplan-Meier method. The percentage of subjects achieving a sCR, CR, VGPR or PR, will be tabulated, and the sCR+CR+VGPR+PR disease rate will be estimated with exact 80% confidence interval. Duration of response among subjects achieving a sCR, CR, VGPR or PR, will be defined as the length of the interval from initial response to progression; duration of response will be tabulated. All toxicities will be tabulated by type and grade.

An interim analysis will be conducted on the first 17 subjects accrued to this trial in order to determine whether the trial should be closed due to insufficient effectiveness. Although 2-year progression-free is the primary endpoint, response (sCR, CR, VGPR, or PR) will be used in the interim analysis as a surrogate endpoint since it can be evaluated much sooner than progression. The response rate of newly diagnosed patients with MM varies across published Phase II and III trials from 40% to 90%. When it becomes obvious that less than 8 of the first 17 subjects on induction therapy will be responders (e.g., if only 3 of the first 13 subjects respond), the study will close.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age 18 years or older at the time of signing the consent.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Multiple myeloma (MM) diagnosed according to the following standard criteria:

   * Monoclonal plasma cells in bone marrow ≥10% and/or presence of biopsy-proven plasmacytoma
   * Monoclonal protein present in serum and/or urine Myeloma-related organ dysfunction (1 or more) (C) Calcium elevation in blood (serum calcium >10.5 mg/L or ULN) (R) Renal insufficiency (SCr >2 mg/dL) (A) Anemia (hemoglobin <10 g/dL or 2g <normal) (B) Lytic bone lesions or osteoporosis
5. Measurable disease requiring systemic therapy.
6. High risk multiple myeloma defined by the presence of one or more of the following:

   * Deletion of chromosome 13 by metaphase analysis (standard cytogenetics)
   * deletion of 17p13 (p53) by Fluorescence in situ hybridization (FISH) or metaphase analysis
   * t(4;14) by FISH
   * t(14;16) by FISH
   * t(8;14) by FISH
   * t(14;20) by FISH
   * hypodiploidy detected by FISH or metaphase analysis
   * any complex cytogenetic abnormality detected by metaphase analysis, with the exception of hyperdiploidy
7. No previous treatment with systemic therapy or radiation therapy lasting more than 4 weeks duration.
8. At least 7 days since date of last radiation or systemic treatment for MM.
9. Eastern Cooperative Oncology Group (ECOG) performance status of < or =2 at study entry.(0=Fully active; 1=Restricted but ambulatory; 2=Ambulatory but unable to work)
10. All study participants must be registered into the mandatory RevAssist® program, and willing and able to comply with the requirements.
11. Females of childbearing potential (FCBP) must have negative pregnancy test with a sensitivity of >/=50 milli-International unit (mIU)/mL within 10-14 days prior to and within 24 hours of prescribing lenalidomide and must use 2 acceptable methods of birth control, one highly effective method and one other effective method AT THE SAME TIME, >4 weeks before taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree not to father a child and agree to use a latex condom even if he has had a successful vasectomy, if partner is FCBP.
12. Disease free of prior malignancies for >5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast
13. Able to take 325 mg aspirin daily as prophylactic anticoagulation for the duration of protocol therapy.
14. Receive concomitant therapy with bisphosphonates if bony lesions are present at time of enrollment.

Exclusion criteria

1. Any serious medical condition, laboratory abnormality, or psychiatric illness to prevent the subject from signing the consent.
2. Pregnant or breast feeding females.
3. Any condition which places the subject at unacceptable risk or confounds the ability to interpret data from the study.
4. Abnormal laboratory test results within these ranges:

   * Absolute neutrophil count < 1.0 x 109/L
   * Platelet count < 50 x 109/L (Subjects with severe pancytopenia (not meeting the above criteria) due to myeloma involvement of > 70% bone marrow are eligible)
   * Serum creatinine > 2.5 mg/dL or ≥ 3.0 mg/dL if due to multiple myeloma.
   * Total bilirubin > 2.0 mg/dl
5. History of allergy to any of the study medications, their analogues, or excipients in the various formulations
6. Concurrent use of other anti-cancer agents or treatments.
7. Known HIV positivity
8. Known Active Hepatitis A, B or C
9. Erythema nodosum characterized by a desquamating rash while taking thalidomide or similar drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-08; Primary Completion 2012-12 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Gasparetto, MD, Principal Investigator — Duke University; David Hurd, MD, Principal Investigator — Wake Forest University Health Sciences; Peter M Voorhees, MD, Principal Investigator — UNC Hospitals, University of North Carolina - Chapel Hill; Jeffrey A. Zonder, MD, Principal Investigator — Karmanos Cancer Center, Wayne State University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in July, 2008 and ended in October, 2010. Subjects were identified from Duke University Medical Center Hematologic Malignancies and Cellular Therapy program and University of North Carolina at Chapel Hill Lineberger Cancer Center for all demographic groups who meet the eligibility criteria.
Groups:
- High-risk Multiple Myeloma: Lenalidomide Induction (with Low Dose Dexamethasone) Therapy Followed by Low Dose Melphalan, Prednisone, Lenalidomide and Bortezomib Sequential Maintenance Therapy
  Lenalidomide Induction: Induction: Lenalidomide 25 mg daily on Days 1-21 followed by 7 day rest and Dexamethasone 40 mg by mouth (po) daily on Days 1, 8, 15 and 22 every 28 days for 4 cycles.
  Sequential Maintenance Therapy: Subjects who achieve >partial response (PR) following induction therapy will receive repeating triplet cycles of alternating low dose therapy until progression, poor tolerance or toxicity. Subjects who complete 24 months of maintenance will be removed from study unless they achieved > stable disease (SD) from maintenance (per discussion with physician):
  * 325 mg aspirin for deep vein thrombosis (DVT) prophylaxis
  * Cycle 1, 4, 7, etc. - bortezomib 1.3 mg/m2 on day 1 and 8 of a 28-day cycle
  * Cycle 2, 5, 8 etc. - Melphalan 6 mg/m2 by mouth (po) daily on Days 1-7
  * Prednisone 60 mg /m2 po daily on
Period: Induction Therapy
Arm/Group | High-risk Multiple Myeloma
Started | 18
Completed | 16
Not Completed | 2
Not completed — Disease Progression | 1
Not completed — Active Hepatitis | 1
Period: Two Years of Maintenance Therapy
Arm/Group | High-risk Multiple Myeloma
Started | 16
Completed | 3
Not Completed | 13
Not completed — Disease Progression | 8
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Subjects enrolled and able to initiate induction therapy.
Groups:
- High-risk Multiple Myeloma: Lenalidomide Induction (with Low Dose Dexamethasone) Therapy Followed by Low Dose Melphalan, Prednisone, Lenalidomide and Bortezomib Sequential Maintenance Therapy
  Induction: Lenalidomide 25 mg daily on Days 1-21 followed by 7 day rest and Dexamethasone 40 mg by mouth (po) daily on Days 1, 8, 15 and 22 every 28 days for 4 cycles.
  Maintenance Therapy: Subjects who achieve >partial response (PR) after induction will receive repeating triplet 28-day cycles of alternating low dose therapy until progression, poor tolerance or toxicity. Subjects who complete 24 months of maintenance will be removed from study unless they achieved > stable disease (SD) from maintenance:
  * 325 mg aspirin for deep vein thrombosis (DVT) prophylaxis
  * Cycle 1, 4, 7, etc. - bortezomib 1.3 mg/m2 on day 1 and 8
  * Cycle 2, 5, 8 etc. - Melphalan 6 mg/m2 by mouth (po) daily on Days 1-7
  * Prednisone 60 mg /m2 po daily on Days 1-7
  * Cycle 3, 6, 9, etc. Lenalidomide 10 mg po daily on Days 1-21.
Arm/Group | High-risk Multiple Myeloma
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 9
  More than one race | 0
  Unknown or Not Reported | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival (PFS) is defined for all subjects as the time from the date of initiation of treatment to the date of first documentation of relapse, progression, or death due to any cause. Full restaging was performed at 6, 12, 18, 24, 36, 48, 60, 72 months). PFS survival will be estimated and plotted with the Kaplan-Meier method. The median will be calculated with 95% confidence intervals.
Time Frame: 2 years
Population: Subjects enrolled and able to initiate induction therapy.
Measure: Number; unit: participants
Arm/Group | High-risk Multiple Myeloma
Number analyzed (Participants) | 18
participants
  PFS at 2 years | 3
  PFS at 1 year | 9

2. Secondary Outcome: Time to Response
Description: Time to response will be measured in the population of subjects with a confirmed response as the time from the date of initiation of treatment to the date of the first documentation of a confirmed response. Full restaging was performed at 6, 12, 18, 24, 36, 48, 60, 72 months). Time to response will be estimated and plotted with the Kaplan-Meier method. The median will be calculated with 95% confidence intervals.
Time Frame: 6 months
Population: Subjects who responded to drug induction therapy.
Measure: Mean (Full Range); unit: months
Arm/Group | High-risk Multiple Myeloma
Number analyzed (Participants) | 16
months | 2 [1.5 to 5]

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the date of initiation of treatment to the date of death due to any cause. Overall response rate will be estimated with its 80% confidence interval, and the numbers of subjects achieving a sustained complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), or stable disease (SD) will be tabulated. Overall survival will be estimated and plotted with the Kaplan-Meier method. The median will be calculated with 95% confidence intervals.
Time Frame: 6 years
Population: Subjects who initiated drug therapy. Eleven patients are still alive as of 2/28/14.
Measure: Mean (Full Range); unit: months
Arm/Group | High-risk Multiple Myeloma
Number analyzed (Participants) | 18
months | 36 [4 to 54]

4. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) is defined for all patients as the time from initiation of treatment to disease progression with deaths owing to causes other than progression not counted as events, but censored (Durie et al., 2006).
Time Frame: 6 years
Population: Subjects who experienced disease progression.
Measure: Mean (Full Range); unit: months
Arm/Group | High-risk Multiple Myeloma
Number analyzed (Participants) | 12
months | 11 [2 to 27]

5. Secondary Outcome: Duration of Response
Description: The duration of response, defined only among the responders, is measured from start of achieving Partial Response (PR) [first observation of PR before confirmation] to the time of disease progression, with deaths owing to causes other than progression not counted as events, but censored (Durie et al., 2006). Duration of response will be estimated and plotted with the Kaplan-Meier method. The median will be calculated with 95% confidence intervals.
Time Frame: 6 years
Measure: Mean (Full Range); unit: months
Arm/Group | High-risk Multiple Myeloma
Number analyzed (Participants) | 16
months | 11 [1 to 25]

ADVERSE EVENTS:
Time Frame: Monitoring of adverse events was conducted through the study period and 30 days following the last dose of lenalidomide. All subjects with adverse events were monitored until resolved or determined to be due to a subject's intercurrent illness.
Description: Toxicities and adverse events were scored using National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. The investigator evaluated each adverse experience for its relationship to the test drug and for its seriousness.
Arm/Group | High-risk Multiple Myeloma
Serious Adverse Events (participants affected / at risk) | 4/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-risk Multiple Myeloma (N=18)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Cardiac Ischemia / infarction (Cardiac disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Acute Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1) — Bacteremia
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Muscular / skeletal hypoplasia (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) — fainting
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) — Back Pain
Pain - Other (General disorders) | 2 (2) — Abdominal Pain
Thrombosis / thrombus / embolism (Vascular disorders) | 1 (1) — Deep Vein Thrombosis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-risk Multiple Myeloma (N=18)
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 1 (1)
thrombosis (Blood and lymphatic system disorders) | 1 (1)
Bacteremia (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5)
anemia (Blood and lymphatic system disorders) | 10 (10)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 15 (15)
leukopenia (Blood and lymphatic system disorders) | 10 (10)
Lymphopenia (Blood and lymphatic system disorders) | 13 (13)
Lymphocytopenia (Blood and lymphatic system disorders) | 4 (4)
Neutrophils / granulocytes (ANC / AGC) (Blood and lymphatic system disorders) | 18 (20)
Platelets (Blood and lymphatic system disorders) | 12 (12)
thrombocytopenia (Blood and lymphatic system disorders) | 9 (9)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Cardiac Left Ventricular Function (Cardiac disorders) | 1 (1)
Constitutional Symptoms - Other (Specify, __) (General disorders) | 1 (1)
Decreased Libido (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 15 (15)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 10 (10)
Insomnia (General disorders) | 10 (10)
Rigors / chills (General disorders) | 4 (4)
Sweating (diaphoresis) (General disorders) | 1 (1)
Weight gain (General disorders) | 3 (3)
Weight loss (General disorders) | 1 (1)
Dermatology / Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 1 (1)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cold sore - left upper lip (Skin and subcutaneous tissue disorders) | 1 (1)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Excoriation bilateral dorsal aspect of feet, related to scratching (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperpigmentation - nailbeds (Skin and subcutaneous tissue disorders) | 1 (1)
Induration, CS (Skin and subcutaneous tissue disorders) | 1 (1)
Peeling skin, intermittent, NCS (Skin and subcutaneous tissue disorders) | 1 (1)
Redness-feet (Skin and subcutaneous tissue disorders) | 1 (1)
Right ankle erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3)
Hair Loss / Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus / itching (Skin and subcutaneous tissue disorders) | 8 (8)
Rash / desquamation (Skin and subcutaneous tissue disorders) | 13 (13)
Hot flashes / flushes (Endocrine disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 8 (8)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 11 (11)
Bleeding (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Heartburn / dyspepsia (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 10 (10)
Taste Alteration (dysgeusia) (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (5)
Hemorrhage / Bleeding - Other (Specify, __) (Blood and lymphatic system disorders) | 2 (2)
Infection - Other (Cellulitis) (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 9 (9)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 5 (5)
Edema (Blood and lymphatic system disorders) | 18 (19)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 4 (4)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 4 (4)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 7 (7)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 6 (6)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 (3)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Decreased Neutrophils (Metabolism and nutrition disorders) | 1 (1)
Uric Acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint-function (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 5 (5)
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Parasthesias (Nervous system disorders) | 1 (1)
Mood Swings (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 2 (2)
Confusion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4)
Mood Alteration - Anxiety (Nervous system disorders) | 6 (6)
Mood Alteration - Depression (Nervous system disorders) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 10 (10)
Syncope (fainting) (Nervous system disorders) | 5 (5)
Tremor (Nervous system disorders) | 2 (2)
Dry Eye Syndrome (Eye disorders) | 2 (2)
Ocular / Visual - Other (Specify, __) (Eye disorders) | 1 (1)
Vision - blurred vision (Eye disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 18 (33)
Pain - General (Nervous system disorders) | 4 (4)
Pain - Head / headache (Eye disorders) | 1 (1)
Pain - Other (Specify, __) (Eye disorders) | 1 (1)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cyanosis of toes (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis / pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary / Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Renal / Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 1 (1)
Malodorous urine (Renal and urinary disorders) | 1 (1)
Urinary frequency / urgency (Renal and urinary disorders) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 2 (2)
Dry mouth (General disorders) | 1 (1)
Early satiety, CS (General disorders) | 1 (1)
Esophageal spasms (General disorders) | 1 (1)
Food Aversions, CS (General disorders) | 1 (1)
Hiccups (General disorders) | 1 (1)
Increased thirst (General disorders) | 1 (1)
Oral lesion (General disorders) | 1 (1)
Bilateral facial swelling (General disorders) | 1 (1)
Paresthesias- Intermittent (General disorders) | 1 (1)
Right Breast Pressure (General disorders) | 1 (1)
Sore throat intermittent (General disorders) | 2 (2)
Sternal Discomfort (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes